CLINICAL TRIAL: NCT01930084
Title: ENGAGE4HEALTH: A Combination Strategy for Linkage and Retention in HIV Care Among Adults in Mozambique
Brief Title: ENGAGE4HEALTH: A Combination Intervention Strategy for Linkage and Retention in Mozambique
Acronym: E4H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Batya Elul, Assistant Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAL1354; USAID-OAA-A-12-00027 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: HIV
Keywords: HIV; linkage; retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combination intervention + incentives (Experimental): 1. Point of care CD4+ after HIV diagnosis
  2. Accelerated ART initiation
  3. SMS appointment reminders
  4. Non-cash financial incentives (FI)
  Interventions: Other: Point of care CD4+ after HIV diagnosis; Other: Accelerated ART initiation; Behavioral: SMS appointment reminders; Other: Non-cash Financial Incentives
- Combination intervention strategy(CIS) (Experimental): 1. Point of care (POC) CD4+ after HIV diagnosis
  2. Accelerated ART initiation
  3. SMS appointment reminders
  Interventions: Other: Point of care CD4+ after HIV diagnosis; Other: Accelerated ART initiation; Behavioral: SMS appointment reminders
- Standard of care (SOC) (No Intervention): Standard of care, no intervention

INTERVENTIONS:
Other: Point of care CD4+ after HIV diagnosis — Point of care (POC) CD4+ testing immediately following HIV diagnosis
  Arms: Combination intervention + incentives; Combination intervention strategy(CIS)
Other: Accelerated ART initiation — Accelerated ART initiation for eligible participants delivered by facility personnel
  Arms: Combination intervention + incentives; Combination intervention strategy(CIS)
Behavioral: SMS appointment reminders — Cellular appointment reminders delivered by study personnel
  Arms: Combination intervention + incentives; Combination intervention strategy(CIS)
Other: Non-cash Financial Incentives — Non-cash Financial Incentives
  Arms: Combination intervention + incentives

SUMMARY:
Purpose: To compare the effectiveness of a combination intervention strategy (CIS), consisting of point of care (POC) CD4+ testing immediately following HIV diagnosis and accelerated ART initiation for eligible participants delivered by facility personnel, and cellular appointment reminders delivered by study personnel, to the standard of care (SOC) on linkage to and retention in HIV care at 12 months among adults testing positive for HIV in Mozambique. Additionally, the protocol will assess the incremental effectiveness of CIS+ non-cash financial incentives (FI) compared to CIS without FI on study outcomes.

DETAILED DESCRIPTION:
Design: Two-arm cluster site-randomized trial with a pre-post intervention two-sample design nested in the intervention arm.

Study Population: The study population is any adult who tests HIV positive at the HIV counseling and testing points participating in this study. The study unit (SU), the level of randomization for the study, includes specific HIV counseling and testing points at primary health care clinics and the HIV care and treatment services located in the same health facility. A total of 10 SU will be included.

Sample Size: A total of 2,250 adults from the 10 study units will be included in the study, 750 in the SOC arm, 750 receiving CIS without FI and 750 receiving CIS+FI.

Participants will be enrolled and followed for 12 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Testing HIV positive at the largest-volume HIV point of testing (other than prevention of mother-to-child transmission or tuberculosis) at SU with written proof of test result
* Agreeing to be referred to the HIV care services associated with the SU
* Agreeing to provide locator information
* Agreeing to adhere to study procedures, including a baseline interview, interviews 1 and 12 months after study enrollment, and extraction of data from the HIV care and treatment electronic database
* Able to provide informed consent

Exclusion Criteria:

* Being pregnant at study enrollment
* Planning on leaving the community where they currently reside in the next 12 months
* Enrolled in HIV care in the past 6 months at any clinic
* Initiated ART (for any duration) in the past 6 months at any clinic
* Currently on ART
* Does not speak or understand Portuguese or Xitswa/Matswa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2004 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Linkage to HIV care within 1 month of HIV testing and retention in care 12 months after testing. | 1 month and 12 months after testing
  An increase in linkage to HIV care within 1 month of HIV testing and retention in care 12 months after testing. Participants are considered to achieve this outcome if they successfully link to the SU HIV care services within 1 month of testing HIV positive as measured from the electronic patient-level database used at the HIV care clinic (EPTS).

SECONDARY OUTCOMES:
Time to linkage to care | 12 months
  A decrease in the median time to linkage to care

OTHER OUTCOMES:
Time from ART eligibility to ART initiation | 12 months
Proportion of participants with new WHO Stage III/IV event or hospitalization | 12 months
Mortality rate 12 months after HIV diagnosis | 12 months
Costs and incremental cost-effectiveness ratio of CIS and of CIS+FI | 12 months
Proportion of patients receiving POC CD4+ test, short message service (SMS) reminders, accelerated ART initiation (among those eligible based on POC CD4+ test result), and FI | 12 months
Proportion of patients reporting that interventions were highly acceptable | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Batya Elul, PhD, MSc, Principal Investigator — Columbia University
Locations (10):
- Mozambique (10):
  - Chicuque Health Center, Inhambane
  - Massinga Health Center, Inhambane
  - Maxixe Health Center, Inhambane
  - Morrumbene Health Center, Inhambane
  - Urbano Health Center, Inhambane
  - Zavala Health Center and Inharrime Health Center, Inhambane
  - Bagamoio Health Center, Maputo
  - Jose Macamo Health Center, Maputo
  - Mavalane General Hospital, Maputo
  - Zimpeto Health Center, Maputo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elul B, Lamb MR, Lahuerta M, Abacassamo F, Ahoua L, Kujawski SA, Tomo M, Jani I. A combination intervention strategy to improve linkage to and retention in HIV care following diagnosis in Mozambique: A cluster-randomized study. PLoS Med. 2017 Nov 14;14(11):e1002433. doi: 10.1371/journal.pmed.1002433. eCollection 2017 Nov. PMID 29136001
- [Derived] Sutton R, Lahuerta M, Abacassamo F, Ahoua L, Tomo M, Lamb MR, Elul B. Feasibility and Acceptability of Health Communication Interventions Within a Combination Intervention Strategy for Improving Linkage and Retention in HIV Care in Mozambique. J Acquir Immune Defic Syndr. 2017 Jan 1;74 Suppl 1(Suppl 1):S29-S36. doi: 10.1097/QAI.0000000000001208. PMID 27930609
- [Derived] Elul B, Lahuerta M, Abacassamo F, Lamb MR, Ahoua L, McNairy ML, Tomo M, Horowitz D, Sutton R, Mussa A, Gurr D, Jani I. A combination strategy for enhancing linkage to and retention in HIV care among adults newly diagnosed with HIV in Mozambique: study protocol for a site-randomized implementation science study. BMC Infect Dis. 2014 Oct 15;14:549. doi: 10.1186/s12879-014-0549-5. PMID 25311998